CLINICAL TRIAL: NCT04322045
Title: A Clinical Study on the Efficiency of Prostate Cancer Screening by the Combination of Serum PSA Assay，Multi-parametric MRI and Targeted Prostate Biopsy Among Males in Nanjing
Brief Title: Combined Prostate-specific Antigen, Multi-parametric MRI and Targeted Prostate Biopsy for Prostate Cancer Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Executive officer of Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IUNU-PC-102
Record Dates: First submitted 2020-01-27; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants (Experimental): All tested serum PSA. Some conducted mpMRI with/without prostate biopsy under instruction.
  Interventions: Diagnostic Test: multi-parametric MRI

INTERVENTIONS:
Diagnostic Test: multi-parametric MRI — Multi-parametric MRI will be suggested for those PSA ≥4 ng/mL, PI-RADS v2 score will be used to evaluate images.
  Other Names: targeted prostate biopsy

SUMMARY:
The study aims to investigate the incidence of prostate cancer among males in Nanjing and whether a combination of PSA, multi-parametric MRI and targeted biopsy is a feasible approach for screening prostate cancer in China.

DETAILED DESCRIPTION:
The investigators are going to collect serum samples and clinical information from men aged ≥50 years taking physical examination in community health service centers in Nanjing. The investigators will propose mpMRI for those with serum PSA ≥4 ng/mL. Transperineal systematic biopsy (TPSB) combined with MRI /ultrasound fusion targeted biopsy (TB) will be offered for those scored ≥3 on the Prostate Imaging-Reporting and Data System Version 2 (PI-RADS v2). TPSB alone will be offered for those scored <3 and serum PSA ≥10 ng/mL. Subjects with serum PSA between 4 ng/mL and 10 ng/mL and PI-RADS score <3 points will be referred to follow-up examinations every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50
* (Eastern Cooperative Oncology Group)ECOG grade: 0-1
* Normal organic function indexes:
* (absolute neutrophil count)ANC ≧1.5×109/L
* (platelet count)PLT ≧100×109/L
* Hb ≧90 g/L
* (total bilirubin)TBIL ≦1.5×ULN
* (aspartate aminotransferase)ALT≦2.5×ULN
* (alanine aminotransferase)AST ≦2.5×ULN
* (blood urea nitrogen)BUN (orUREA) and Cr ≦1.5×ULN

Exclusion Criteria:

* Former serum PSA detection
* Having took Proscar in the past 3 months
* Suffered from any other malignant tumor in the past 5 years
* History of acute urinary retention, acute or chronic bacterial or abacterial prostatitis within 6 weeks or other recent infection of the urinary system
* Having took Proscar in the past 3 months
* Suffered from any other malignant tumor in the past 5 years
* History of acute urinary retention, acute or chronic bacterial or abacterial prostatitis within 6 weeks or other recent infection of the urinary system

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Screening for prostate cancer is conducted only among males
Enrollment: 10000 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of prostate cancer | 3 years
  Incidence of prostate cancer among males ≥50 years old

SECONDARY OUTCOMES:
Number of participants with different gleason scores | 3 years
  Gleason score of prostate cancer patients, Including 7 degrees:3+3=6,3+4=7,4+3=7,4+4=8,4+5=9,5+4=9,5+5=10.
Number of participants with different clinical stages | 3 years
  Clinical stage of prostate cancer patients according to the eighth version of American Joint Committee on Cancer(AJCC) guideline for prostate cancer.
Number of participants with different risk groups | 3 years
  Devided to three risk groups(high-medium-low) according to D'Amico risk groups of prostate cancer.
Number of participants with different prognostic stage groups | 3 years
  Prognostic stage of prostate cancer patients according to the eighth version of American Joint Committee on Cancer(AJCC) guideline for prostate cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
not willing to share